CLINICAL TRIAL: NCT01124734
Title: Phase II Trial of High Dose Interleukin-2 Followed by Intermittent Low Dose Temozolomide in Patients With Metastatic Malignant Melanoma
Brief Title: High Dose Interleukin-2 Followed by Intermittent Low Dose Temozolomide in Patients With Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Joseph Drabick, Professor of Medicine, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSHCI 09-067
Record Dates: First submitted 2010-03-04; First posted 2010-05-17 (Estimated); Results first posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-01

CONDITIONS: Malignant Melanoma
Keywords: Metastatic melanoma
MeSH Terms: conditions — Melanoma | interventions — Interleukin-2; Temozolomide

STUDY DESIGN:
Intervention Model Description: Single group, open label study
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Course 1 Cycle 1 and Cycle 2 (Experimental): Course 1 Cycle 1: Participants will be given high-dose Interleukin-2 (HD IL-2) 600,000 IU/kg, up to 14 doses at 8 hour intervals.
  Course 1 Cycle 2: Participants will be given high-dose Interleukin-2 (HD IL-2) 600,000 IU/kg, up to 14 doses at 8 hour intervals. On the day after discharge, patients will be given oral temozolomide at 75 mg/m2 daily for 21 days.
  Interventions: Drug: Interleukin-2; Drug: Temozolomide

INTERVENTIONS:
Drug: Interleukin-2 — Participants will receive IL-2 up to a maximum of 14 doses at 600,000 IU/kg
  Other Names: IL-2
Drug: Temozolomide — Participants receive temozolomide at 75 mg/m2 after completion of the second cycle of high dose IL-2. Participants take the medication at bedtime daily. Four weeks after Cycle 2 of a course, they would take it for 21 days.
  Other Names: Temodar, Temodal, Temcad; Temodal

SUMMARY:
The investigators have observed that many patients who had received high dose Interleukin-2 (IL2) and failed to respond to it but who then go immediately to temozolomide seemed to enjoy extremely good responses which seem better quality and longer duration than typically observed for temozolomide alone. To date, the investigators have observed 5 sequentially treated patients with metastatic melanoma who had failed high dose IL-2 but who then went on to receive immediate temozolomide. Two of these patients had complete responses and 3 had very strong partial response. In a recent phase II study of extended low dose temozolomide alone given in the same manner as the post IL-2 patients noted above, the response rate was 12.5% and all of these were partial responses only. The responses that the investigators observed were at a much higher rate of response as well as much better quality than expected for temozolomide. The responses were also better than those observed when temozolomide was given first and then followed by high dose IL-2. The investigators concluded that perhaps the major benefit the investigators observed was a result of the prior high dose IL-2 therapy modulated by the temozolomide and that the sequence of treatment was clearly crucial for this response.

DETAILED DESCRIPTION:
Metastatic malignant melanoma remains a disease with a very poor prognosis and median survival duration of less than one year. Durable remissions with conventional therapy are rare and therefore clinical trials remain a primary treatment modality for metastatic disease. There are 2 currently FDA-approved therapies for metastatic melanoma. Chemotherapy with single agent parenteral dacarbazine or its oral pro-drug, temozolomide, are capable of producing responses in 6.5 to 20% of patients. These responses are usually minor to partial at best and are not durable. Combination with other chemotherapeutic drugs has not been successful. The immune system also seems to play a role in malignant melanoma. High dose Interferon therapy is the current standard therapy for the adjuvant treatment of stage IIB, IIC and III melanoma after surgical resection in which it has shown to result in modest improvements in disease free survival and overall survival. In metastatic disease, various immunologic approaches have been employed as well. High dose IL-2 can produce a response rate of about 10-15% in patients with metastatic melanoma. About 5-10% of responses are complete and some of these complete responses are durable so that the lucky few patients who have a durable complete response are for all intents and purposes cured. Attempts to combine chemotherapy with immunotherapy, although improving response rates, has not impacted survival as summarized in recent meta-analysis.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed metastatic malignant melanoma
* Age > 18 years
* Eastern Cooperative Oncology Group performance status of 0 or 1
* Patients considered good candidate for conventional high dose IL-2
* No chemotherapy, hormonal therapy, immunotherapy or radiation therapy within 1 month of entry
* Patients with a history or clinical evidence of brain metastasis must have completed radiation therapy or surgical treatment of brain lesions and have no evidence of central nervous system progression for at least 8 weeks at the time of enrollment.
* Patients may have had prior high dose IL-2 or temozolomide but not together or with high dose IL-2 followed by temozolomide
* Patients may have had prior high dose interferon as adjuvant treatment for high risk melanoma
* Serum creatinine < 2 mg/dL
* Bilirubin < 2 mg/dL

Exclusion Criteria:

* Inability to provide informed consent
* Hypersensitivity to temozolomide or HD IL-2
* Active gastrointestinal disorder or cardiac disorders
* Ejection fraction < 50% by echocardiogram or corrected diffusing capacity of lung for carbon monoxide < 50% on diffusion capacity testing pulmonary function tests
* platelets < 100 K, neutrophils < 1000
* Serum Creatinine < 2 x the upper limits of normal
* Chronic use of steroids other than for simple adrenal replacement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-05; Primary Completion 2017-07-18 (Actual); Study Completion 2018-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph J Drabick, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single center study conducted at Penn State Hershey Medical Center Cancer Institute. The study was carried out in the Cancer Institute outpatient clinic. Accrual was initiated 9/07/2011 and completed completed 04/28/2014. Participants remained on study for long term follow up. The study closed in July 2018.
Pre-assignment Details: Participants were excluded if they received any chemotherapy, hormonal therapy, immunotherapy, or radiation therapy within 1 month of entry to the study.
Groups:
- Course 1 Cycle 1 and Cycle 2: This study is a single arm study. All participants received the same treatment regimen.
  For initiation of study intervention (Course 1 - Cycle 1) participants are admitted inpatient for Course 1 Cycle 1 of HD IL-2 treatment. Participants will be given as many doses of IL-2 as tolerated up to a maximum of 14 at 8 hr intervals as allowed by the algorithm at 600,000 IU/kg. Participants will be discharged when the acute toxicities of the IL-2 have subsided.
  Course 1 Cycle 2: After discharge, participants will be reassessed on or about 10 days after discharge (D10) and will be re-admitted to initiate Course 1 Cycle 2. For this Cycle 2, participants will be given as many doses of IL-2 as tolerated up to a maximum of 14 at 8 hr intervals as allowed by the algorithm at 600,000 IU/kg. After completion of this cycle 2 HD IL-2, they would begin Temzolomide at 75 mg/m2 on the day after hospital discharge. Participants will continue with Temzolomide for a total of 21 days.
Period: Overall Study
Arm/Group | Course 1 Cycle 1 and Cycle 2
Started | 17
Completion of Course 1 Cycle 1 | 17 (All 17 participants successfully completed Course 1 Cycle 1)
Initiation of Course 1 Cycle 2 | 17
Completed | 0 (Closed to accrual)
Not Completed | 17
Not completed — Disease progression | 13
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Elected for alternative treatment | 2

BASELINE CHARACTERISTICS:
Population: All participants had melanoma.
Groups:
- Course 1 Cycles 1 and 2: Course 1 Cycles of Part 1: Participants will be given High-Dose Interleukin-2 (HD IL-2) 600,000 IU/kg, up to 14 doses at 8 hour intervals. Interleukin-2: up to a maximum of 14 doses at 600,000 IU/kg
  Course 2: Patients will be given High-Dose Interleukin-2 (HD IL-2) 600,000 IU/kg, up to 14 doses at 8 hour intervals. On the day after discharge, patients will be given oral temozolomide at 75 mg/m2 daily for 21 days. Interleukin-2: up to a maximum of 14 doses at 600,000 IU/kg. Temozolomide: Patients would receive temozolomide at 75 mg/m2 after discharge from receipt of the second cycle of high dose IL-2. Patients would take the medication at bedtime daily. Four weeks after cycle 2 of a course, they would take it for 21 days.
Arm/Group | Course 1 Cycles 1 and 2
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Per NIH defined Racial and Ethnic Categories
  Participants
    Hispanic or Latino | 0
    Not Hispanic or Latino | 17
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants] — Region as defined by Country (i.e. United States, Canada, Vietnam, etc)
  Participants
    United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response to High-Dose Interleukin-2 (H-D IL-2) Followed by Low Dose Temozolomide
Description: Clinical response was measured using the Response Evaluation Criteria In Solid Tumors (RECIST) criteria categorizing responses as complete response (CR), partial response (PR), minor response (MR), stable disease (SD), or progressive disease (PD).
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Groups:
- Course 1 Cycle 1: This study is a single arm study. All participants received the same treatment regimen.
  Participants were given High-Dose Interleukin-2 (HD IL-2) 600,000 IU/kg, up to 14 doses at 8 hour intervals.
  Interleukin-2: up to a maximum of 14 doses at 600,000 IU/kg
- Course 1 Cycle 2: Patients will be given High-Dose Interleukin-2 (HD IL-2) 600,000 IU/kg, up to 14 doses at 8 hour intervals. On the day after discharge, patients will be given oral temozolomide at 75 mg/m2 daily for 21 days.
  Interleukin-2: up to a maximum of 14 doses at 600,000 IU/kg
  Temozolomide: Patients would receive temozolomide at 75 mg/m2 after discharge from receipt of the second cycle of high dose IL-2. Patients would take the medication at bedtime daily. Four weeks after cycle 2 of a course, they would take it for 21 days.
Arm/Group | Course 1 Cycle 1 | Course 1 Cycle 2
Number analyzed (Participants) | 17 | 17
Participants
  Stable Disease | 17 | 4
  Partial Response | 0 | 1
  Progressive Disease | 0 | 9
  Minor Response | 0 | 1
  Complete Response | 0 | 2

2. Primary Outcome: Duration of Response to High-Dose Interleukin-2 (H-D IL-2) Followed by Low Dose Temozolomide
Description: Duration of response is defined as the length (measured in days) from the date of best response to the date of progression (if any), or to the date of last follow-up (if no progression is observed). The duration of response is applicable for those CR/MR/PR/SD subjects only.
Time Frame: 8 years
Population: Duration of response is applicable for those CR/MR/PR/SD subjects only.
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | Course 1 Cycle 1 and Cycle 2
Number analyzed (Participants) | 8
Days | 432.88 [0 to 963.16]

3. Primary Outcome: Safety and Toxicity of H-D IL-2 Followed by Low Dose Temozolomide
Description: Safety and toxicity in this study population was evaluated using the NCI Common Toxicity Criteria. The unit of measure is the number of study participants with one or more unexpected and related (even remotely) SAE.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Course 1 Cycle 1 | Course 1 Cycle 2
Number analyzed (Participants) | 17 | 17
Participants | 0 | 0

4. Secondary Outcome: Effect of High Dose IL2 Followed by Low Dose Temozolomide on Lymphocyte Subsets (Autoimmune Biomarkers)
Description: The effect outcome is measured by the change in percentage of circulating lymphocyte cells (autoimmune biomarkers) that express the noted phenotype. This percentage change is determined by comparing the values obtained within 7 days of participant going off treatment against the baseline values.
Time Frame: 2 years
Population: Of the 17 qualifying participants, 9 underwent baseline (pre-Course 1) testing. Eleven participants consented to and underwent this POST off- treatment testing. Two of the participants tested at Post treatment did not have baseline testing done.
Measure: Mean (Standard Deviation); unit: Percentage of Cells
Groups:
- % of Cells Expressing Phenotype Pre-treatment (BASELINE): % of lymphocyte subset cells (particularly the T-reg cells, on cytokine production and anti-melanoma specific t-cell immune cells) that express the particular phenotype noted. Measured at pre-treatment time period (i.e. baseline)
- % of Cells Expressing Phenotype Within 7 Days of Off-treatment: % of lymphocyte subset cells (particularly the T-reg cells, on cytokine production and anti-melanoma specific t-cell immune cells) that express the particular phenotype noted. Measured within 7 days the participant went off treatment. Note: Off treatment day will vary by participant and response to treatment/other intervening factors (toxicity, withdrawal of IC, etc).
Arm/Group | % of Cells Expressing Phenotype Pre-treatment (BASELINE) | % of Cells Expressing Phenotype Within 7 Days of Off-treatment
Number analyzed (Participants) | 9 | 11
Percentage of Cells
  %CCR7- CD45RO+ of CD4+ Effector Memory | .36 (.10) | .36 (.10)
  %CCR7- CD45RO+ of CD8+ Effector Memory | .31 (.10) | .34 (.16)
  %CCR7- CD45RO- of CD4+ Effector Memory RA+ | .09 (.08) | .08 (.07)
  %CCR7- CD45RO- of CD8+ Effector Memory RA+ | .46 (.18) | .40 (.15)
  %CD25+FoxP3+ of CD4+ (Tregs) | .10 (.05) | .09 (.05)

ADVERSE EVENTS:
Time Frame: Participants were followed for all AEs (Grade 0-V) from enrollment (signing consent) to the day they were rendered off study. The follow up period was indefinite as when off treatment, all were followed for disease status. Total time period for those who remained on study until the end is 8 years.
Description: Definition and processes the same as clinicaltrials.gov terminology.
Arm/Group | Course 1 Cycle 1 | Course 1 Cycle 2
All-Cause Mortality (participants affected / at risk) | 0/17 | 9/17
Serious Adverse Events (participants affected / at risk) | 1/17 | 1/17
Other Adverse Events (participants affected / at risk) | 17/17 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Course 1 Cycle 1 (N=17) | Course 1 Cycle 2 (N=17)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) — Stroke
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) — sinus tachycardia left bundle branch block
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Course 1 Cycle 1 (N=17) | Course 1 Cycle 2 (N=17)
Hyperbilirubinemia (Hepatobiliary disorders) | 6 (20) | 1 (2)
Capillary leak syndrome (Vascular disorders) | 10 (18) | 4 (6) — Capillary leak syndrome
Diarrhea (Gastrointestinal disorders) | 9 (24) | 4 (7)
Mucositis (Gastrointestinal disorders) | 6 (15) | 2 (4)
Flu like symptoms (General disorders) | 9 (18) | 3 (9)
Fatigue (General disorders) | 9 (15) | 2 (2)
Abdominal cramping (Gastrointestinal disorders) | 2 (2) | 0 (0) — Abdominal cramping
Alkaline phosphatase increase (Hepatobiliary disorders) | 5 (8) | 1 (1) — Alkaline phosphatase increase
Alanine aminotransferase increased (Hepatobiliary disorders) | 6 (8) | 1 (2) — Alanine aminotransferase increased
Anemia (Blood and lymphatic system disorders) | 7 (17) | 3 (8) — Anemia
Loss of Appetite - Anorexia (Gastrointestinal disorders) | 6 (10) | 3 (3)
Aspartate aminotransferase increased (Hepatobiliary disorders) | 4 (7) | 2 (2) — Aspartate aminotransferase increased
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) — Back pain
Constipation (Gastrointestinal disorders) | 3 (4) | 0 (0)
Increased creatinine (Renal and urinary disorders) | 6 (11) | 3 (7)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 8 (8) | 3 (3)
Dysgeusia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (10) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 4 (7) | 2 (2)
Hypoalbuminemia (Hepatobiliary disorders) | 7 (15) | 3 (10)
Hypernatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 9 (32) | 3 (9)
Hypokalemia (Metabolism and nutrition disorders) | 4 (7) | 2 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 7 (14) | 3 (6)
Hyponatremia (Metabolism and nutrition disorders) | 6 (15) | 3 (6)
Hypophosphatemia (Metabolism and nutrition disorders) | 8 (18) | 4 (7)
INR increased (Blood and lymphatic system disorders) | 5 (9) | 2 (2)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 4 (8) | 3 (4)
Nausea (Gastrointestinal disorders) | 9 (17) | 3 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 5 (7) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Activated partial thromboplastin time prolonged (Blood and lymphatic system disorders) | 3 (4) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 2 (3) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (24) | 3 (12)
Vomiting (Gastrointestinal disorders) | 7 (14) | 3 (6)
White blood cell decreased (Blood and lymphatic system disorders) | 3 (8) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-09-24): https://cdn.clinicaltrials.gov/large-docs/34/NCT01124734/Prot_SAP_000.pdf